CLINICAL TRIAL: NCT03865160
Title: Low-dose Atropine for Myopia Control in Children, a Prospective, Double-blind, Placebo-controlled, Multicentric, Randomized Clinical Trial
Brief Title: Low-dose Atropine for Myopia Control in Children
Acronym: AIM
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Eye Hospital, Freiburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P001307; DRKS00023337 (Registry Identifier: German Clinical Trials Register (DRKS)); 2020-001575-33 (EudraCT Number)
Record Dates: First submitted 2019-03-03; First posted 2019-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Myopia, Progressive
Keywords: Myopia; Children; Atropine; Low-dose; 0.01; 0.02
MeSH Terms: conditions — Myopia, Degenerative; Myopia | interventions — Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: Year one: arm A atropine 0.02% / arm B placebo Year two: arm A atropine 0.02% / arm B atropine 0.01% Year three: arm A placebo/ arm B atropine 0.01%
Who Masked: Participant, Investigator
Masking Description: Code labelled eye drop containers Blinded investigators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A, Interventional group (Experimental): Treatment period 1: Atropine eye drops, 0.02%, 1 drop/eye, daily for 12 months Treatment period 2: Atropine eye drops, 0.02%, 1 drop/eye, daily for 12 months Treatment period 3: Placebo (NaCl 0.9%) eye drops, 1 drop/eye, daily for 12 months
  Interventions: Drug: Atropine eye drops, 0.02%; Drug: Placebo (NaCl 0.9%) eye drops
- Arm B, Control group (Experimental): Treatment period 1: Placebo (NaCl 0.9%) eye drops, 1 drop/eye, daily for 12 months Treatment period 2: Atropine eye drops, 0.01%, 1 drop/eye, daily for 12 months Treatment period 3: Atropine eye drops, 0.01%, 1 drop/eye, daily for 12 months
  Interventions: Drug: Atropine eye drops, 0.01%; Drug: Placebo (NaCl 0.9%) eye drops

INTERVENTIONS:
Drug: Atropine eye drops, 0.01% — One drop of the above mentioned drug will be installed into each eye daily at bedtime.
  Arms: Arm B, Control group
Drug: Atropine eye drops, 0.02% — One drop of the above mentioned drug will be installed into each eye daily at bedtime.
  Arms: Arm A, Interventional group
Drug: Placebo (NaCl 0.9%) eye drops — One drop of the above mentioned drug will be installed into each eye daily at bedtime.

SUMMARY:
Myopia (nearsightedness) is the most common eye disorder. Only second to age, it is the main risk factor for major degenerative eye diseases such as glaucoma, macular degeneration or retinal detachment. Their risk increases with the degree of myopia. Hence, prevention of myopia and slowing its progression is of high relevance. Almost all clinical studies, including two large randomised clinical trials (RCT) were performed in Asia with Asian study participants. The results indicate that atropine eye drops can attenuate myopic progression in children, even in low concentrations thus minimizing unwanted side effects. However, the cumulative evidence is yet not strong enough to recommend their unrestricted use, especially in a Non-Asian population. We therefore intend to set up an adequately powered RCT comparing atropine 0.02% eye drops with placebo to validate previous findings and to test whether this therapeutic concept holds its promise in a European population.

DETAILED DESCRIPTION:
Myopia (nearsightedness) is the most common developmental eye disorder in the first decades of life. It is the biggest risk factor for sight threatening degenerative eye diseases later in life, second only to age. Its prevalence is increasing worldwide in pandemic dimensions affecting now > 80% in Asian and > 40% in Caucasian populations. Myopia is one of the five eye diseases identified as immediate priorities by the WHO's global initiative for the elimination of avoidable blindness. It usually develops during primary school and its onset and progression are related to environmental factors such as near work and lack of day light exposure, to a lesser degree to genetic factors. Therefore, retardation of myopia progression is a major therapeutic goal. Clinical trials from Asia have shown that 0.01% atropine eye drops can attenuate progression of myopia while inducing only little side effects such as light sensitivity and reduced accommodation. Subsequent data also from Asia have suggested that a concentration of 0.05% atropine is slightly more effective with a still acceptable level of adverse effects. However, it is unclear whether this therapy is equally and sufficiently efficacious in a Caucasian population. It is also unclear which concentration of atropine represents the best compromise between efficacy and safety. Our own uncontrolled pilot data suggest that 0.01% delays progression by about 50% with negligible side effects, but that 0.05% induces a pupil dilation of > 3 mm, which is considered unacceptable. Due to the increasing prevalence also in Europe and an increasing demand from parents for means to retard myopia progression, the trial is the first European large scale randomized clinical trial investigating the safety and efficacy of 0.01% and 0.02% atropine eye drops in comparison to placebo drops. Such a trial is mandatory to substantiate the increasing off-label prescriptions of low-dose atropine in children and to develop clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 8 to 12 years (up to the day before the 13th birthday)
2. Myopia of -1 D to -6 D with reported or documented annual progression ≥ 0.5 D of myopia
3. Written informed consent obtained from patient (if applicable) and parents or legal guardians according to international guidelines and local laws
4. Ability to understand the nature of the trial and the trial related procedures and to comply with them

Exclusion Criteria:

1. Asian or African origin
2. Abnormal binocularity
3. Strabismus
4. Astigmatism >1.5 D
5. Anisometropia >1.5 D
6. History of amblyopia
7. Corrected visual acuity in any eye <0.63
8. Any acquired or developmental organic eye disease
9. Premature birth
10. Any known systemic metabolic disease or chromosomal anomaly
11. Previous use of any kind of contact lenses
12. Previous use of atropine eye drops
13. Epilepsy
14. Known hypersensitivity to the active substances or any of the excipients
15. Participation in any other interventional clinical trial within the last 30 days before the start of this trial
16. Simultaneous participation in other interventional trials which could interfere with this trial; simultaneous participation in registries and diagnostic trials is allowed
17. Contraindications according to the Summary of Product Characteristics (SmPC): Increased intraocular pressure (primary forms of glaucoma or narrow angle glaucoma), chronic rhinitis sicca
18. Caution and pediatric counselling shall be assured if any of the following conditions are present according to the Summary of Product Characteristics (SmPC): Cardiac insufficiency, arrhythmia, coronary stenosis, hyperthyroidism, stomach or bowel stenosis, bowel paralysis, megacolon, muscle weakness, lung edema, hypersensitivity to atropine, spastic paralysis
19. Parents or children with poor understanding of the German language
20. Person who is in a relationship of dependence/employment with the sponsor or the investigator

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Demonstration of superiority of low-dose atropine 0.02% eye drops compared to placebo for myopia control | Baseline - 12 months
  Change in cycloplegic refraction [dioptre (D)/year] after one year will be performed using an analysis of covariance (ANCOVA) model with the annual change in refraction as the dependent variable. The mean value of both eyes is analysed.

SECONDARY OUTCOMES:
Assessment of axial eye length growth under low-dose atropine 0.02% in comparison to placebo | Baseline - 12 months
  Change in axial length [mm/year]. The mean value of both eyes is analysed. Analyses will be performed in a regression model.
Assessment of the categorized rate of change in refraction of low-dose atropine 0.02% compared to placebo | Baseline - 12 months
  The primary endpoint change in cycloplegic refraction after one year will be categorized (patients progressing < 0.25D (dioptre), 0.25D - 0.75D and > 0.75D after one year of treatment) and will be analysed descriptively, giving absolute and relative frequencies of these categories as a supportive analysis.

OTHER OUTCOMES:
Assessment of rebound of myopia progression (refraction) after cessation of atropine 0.02% treatment | 24-months - 36-months
  Change in refraction [D/year] in year 3, to be determined only in the intervention group.
Assessment of rebound of myopia progression (axial length) after cessation of atropine 0.02% treatment | 24-months - 36-months
  Change in axial length [mm/year] in year 3, to be determined only in the intervention group.
Change in refraction [D/year] | intervention group: baseline - 24-months, control group: 12-months - 36-months
  Change in refraction [D/year] after two years of treatment with low-dose atropine 0.02% eye drops (after year 2 in the interventional group) compared to low-dose atropine 0.01% eye drops (after year 3 in the control group).
Change in axial length [mm/year] | intervention group: baseline - 24-months, control group: 12-months - 36-months
  Change in axial length [mm/year] after two years of treatment with low-dose atropine 0.02% eye drops (after year 2 in the interventional group) compared to low-dose atropine 0.01% eye drops (after year 3 in the control group).
Assessment of safety of topical preservative free atropine in comparison to placebo with regard to pupil size | Baseline - 36-months
  Pupil diameter in mm using the IOL Master 500 or 700 or a PlusoptiX device (preferred) at 200 - 300 lux room illumination. Parameter will be listed by site and patient and displayed in summary tables.
Assessment of safety of topical preservative free atropine in comparison to placebo with regard to near vision | Baseline - 36-months
  Visual acuity at near (40 cm distance) using Landolt-C near vision charts (non-crowded version) as decimal acuity. Parameter will be listed by site and patient and displayed in summary tables.
Assessment of safety of topical preservative free atropine in comparison to placebo with regard to accomodation | Baseline - 36-months
  Accommodation in D as the near point by the Royal air force near point rule (RAF) or by the Accommodation Convergence Rule (VISUS GmbH) (mean of three measurements of both eyes). Parameter will be listed by site and patient and displayed in summary tables.
Assessment of safety of topical preservative free atropine in comparison to placebo with regard to pulse rate | Baseline - 36-months
  Pulse rate (per minute): parameter will be listed by site and patient and displayed in summary tables.
Number of participants with treatment-related adverse events as assessed by the current CTCAE v4.0 | Baseline - 36-months
  * A questionnaire about potential side effects will be completed three times during the study course
  * A patient diary of potential side effects will be provided for patients/parents or guardians to complete and bring to each study visit
  * Adverse events will be documented in the eCRF
  The adverse events are displayed in summary tables by treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wolf Lagrèze, Prof., Principal Investigator — Eye Center, Medical Center, University Hospital Freiburg
Locations (19):
- Germany (19):
  - Augen-Zentrum-Nordwest, Augenpraxis Ahaus, Ahaus
  - Universitäts-Augenklinik Bonn, Bonn
  - Uniklinik Köln, Zentrum für Augenheilkunde, Cologne
  - Universitätsklinikum Erlangen, Augenklinik, Erlangen
  - Universitätsklinikum Essen, Klinik für Augenheilkunde, Essen
  - Medical Center - University of Freiburg, Eye Hospital, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Augenklinik, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Klinik und Poliklinik für Augenheilkunde, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Augenheilkunde, Hanover
  - Universitätsklinikum Heidelberg, Augenklinik, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Augenheilkunde, Leipzig
  - Universitätsklinikum Magdeburg A.ö.R., Universitätsaugenklinik, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Augenklinik und Poliklinik, Mainz
  - Ludwig-Maximilians-Universität München, Augenklinik und Poliklinik, München
  - Klinik für Augenheilkunde des UKM, Gebäude D15, Münster
  - Pius-Hospital Oldenburg, Medizinischer Campus Universität Oldenburg, Universitätsklinik für Augenheilkunde, Oldenburg
  - AugenCentrum Rosenheim, Rosenheim
  - Universitätsklinikum Ulm, Klinik für Augenheilkunde, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farassat N, Bohringer D, Kuchlin S, Molnar FE, Schwietering A, Seger D, Hug MJ, Knobel AB, Schneider-Fuchs S, Ihorst G, Wabbels B, Beisse C, Ziemssen F, Schuettauf F, Hedergott A, Ring-Mangold T, Schuart C, Wolf A, Schmickler S, Biermann J, Eberwein P, Hufendiek K, Eckstein A, Gusek-Schneider G, Schittkowski M, Lischka T, Lagreze WA. Low-dose AtropIne for Myopia Control in Children (AIM): protocol for a randomised, controlled, double-blind, multicentre, clinical trial with two parallel arms. BMJ Open. 2023 Apr 20;13(4):e068822. doi: 10.1136/bmjopen-2022-068822. PMID 37080623
- See also: Homepage of AIM (German language) — http://aim-studie.de